CLINICAL TRIAL: NCT00412191
Title: A Pivotal Single-dose Randomised, Parallel-group, Open-label Study to Demonstrate Bioequivalence of 300mg Lamotrigine XR Relative to 100mg + 200mg Lamotrigine XR and to Demonstrate Lack of Food Effect on 300mg Lamotrigine XR in Healthy Male and Female Volunteers
Brief Title: Bioequivalence And Lack Of Food Effects Of 300mg Lamotrigine XR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAM105379
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: healthy volunteers; bioequivalence; food effects
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects in treatment regimen A (Experimental): Subjects in treatment regimen A will receive 100 and 200 mg lamotrigine XR in fasting condition.
  Interventions: Drug: Lamotrigine
- Subjects in treatment regimen B (Experimental): Subjects in treatment regimen B will receive 100 mg lamotrigine XR in fasting condition.
  Interventions: Drug: Lamotrigine
- Subjects in treatment regimen C (Experimental): Subjects in treatment regimen C will receive 100 mg lamotrigine XR in fed condition.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — In treatment regimen A lamotrigine XR tablets will be available 100 and 200mg tablets, for regimen B and C of lamotrigine tablets 300 mg will be available.

SUMMARY:
This study intends to demonstrate bioequivalence and lack of food effect on 300mg lamotrigine XR in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 kg (males) or >45 kg (females) and BMI within the range 19 - 29.9 kg/m2 inclusive.
* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, vital signs and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.

Exclusion Criteria:

* Female subjects of childbearing potential will not be eligible to participate who are unwilling or unable to use an appropriate method of contraception as outlined in the inclusion criteria from at least the commencement of their last normal period prior to the first dose of study medication; and to continue until the first normal period (defined as normal for the woman, both in terms of duration and quantity of menses) after treatment or 5 half lives of the study medication, whichever is the longest.
* Female subject is pregnant (positive serum human chorionic gonadotrophin (hCG) test at screening) or lactating.
* Female subjects using hormonal contraceptive precautions including progesterone-coated IUD
* Female subjects using hormonal replacement therapy.
* Subjects who received lamotrigine in a previous study (subjects who received placebo will be allowed).
* Current smokers of 10 or more cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-02-06 (Actual); Primary Completion 2007-04-27 (Actual); Study Completion 2007-04-27 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics ie Serum lamotrigine Cmax and AUC(0-inf) | taken pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26, 36, 48, 72, 96, 120 and 144 hours following dosing

SECONDARY OUTCOMES:
PK (AUC (0-t), tmax and t1/2 ) | taken pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26, 36, 48, 72, 96, 120 and 144 hours following dosing
safety and tolerability based on physical exam, adverse events, changes in biochemistry, haematology, urinalysis parameters, electrocardiogram parameters, blood pressure and heart rate measure | at Screening, Day -1, Day 1, Day 2 and follow up 7-14 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study LAM105379 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/LAM105379?search=study&search_terms=LAM105379#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM105379 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register